CLINICAL TRIAL: NCT06837948
Title: Neoadjuvant Chemotherapy Combined With Bispecific Antibody Versus Monoclonal Antibody in Locally Advanced Non-Small Cell Lung Cancer: A Multicenter, Randomized Controlled Clinical Trial
Brief Title: Neoadjuvant Chemotherapy Combined With Bispecific Antibody Versus Monoclonal Antibody in Locally Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-026
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — sintilimab; 130-nm albumin-bound paclitaxel; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exploratory arm (Experimental): In this arm, 20 patients with locally advanced Non-small cell lung cancer will receive 4 circles of neoadjuvant PM8002 combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: PM8002; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery
- PM8002 arm (Experimental): Patients with locally advanced Non-small cell lung cancer will be randomized into this arm (70 patients) and receive 4 circles of neoadjuvant PM8002 combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: PM8002; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery
- Sintilimab arm (Active Comparator): Patients with locally advanced Non-small cell lung cancer will be randomized into this arm (70 patients) and receive 4 circles of neoadjuvant Sintilimab combined with platinum-based doublet chemotherapy and those resectable after neoadjuvant therapy will be treated with surgery.
  Interventions: Drug: Sintilimab; Drug: Nab-paclitaxel; Drug: Carboplatin; Procedure: Surgery

INTERVENTIONS:
Drug: PM8002 — Specified dose on specified days.
  Arms: Exploratory arm; PM8002 arm
Drug: Sintilimab — Specified dose on specified days.
  Arms: Sintilimab arm
Drug: Nab-paclitaxel — Specified dose on specified days.
Drug: Carboplatin — Specified dose on specified days.
Procedure: Surgery — Patients with resectable tumor after neoadjuvant therapy will be treated with surgery.

SUMMARY:
Surgical intervention remains the primary treatment option for early-stage lung cancer. With the proven efficacy of immunotherapy in the treatment of advanced non-small cell lung cancer (NSCLC), neoadjuvant immunotherapy has increasingly become a focal point of research. Blocking vascular endothelial growth factor (VEGF) not only inhibits the proliferation of vascular endothelial cells and the formation of new blood vessels but also improves the tumor microenvironment and enhances the infiltration of cytotoxic T lymphocytes within it. Simultaneously targeting the VEGF and PD-L1 pathways can create a synergistic anti-cancer effect. PM8002 injection is a bispecific antibody drug that targets both PD-L1 and VEGF, functioning as a dual-action agent that combines immune suppression and anti-angiogenesis. In patients with locally advanced stage II-III NSCLC, neoadjuvant therapy that concurrently targets PD-L1/VEGF in combination with chemotherapy can improve pathological response rates, provided that the safety of the drug combination is maintained. This approach offers additional benefits to patients, prolongs event-free survival (EFS), and improves prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient shall sign the Informed Consent Form.
2. Aged 18 ≥ years.
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and stage II-III confirmed by imageological examinations (CT, PET-CT or EBUS)，and have not previously received anti-tumor treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1.
5. Life expectancy is at least 12 weeks.
6. At least 1 measurable lesion according to RECIST 1.1.
7. Patients with good function of other main organs (liver, kidney, blood system, etc.)
8. Patients with lung function can tolerate surgery;
9. Without systematic metastasis (including M1a, M1b and M1c);
10. Fertile female patients must voluntarily use effective contraceptives not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later) during the study period, and urine or serum pregnancy test results within 7 days prior to enrollment are negative.
11. Unsterilized male patients must voluntarily use effective contraception during the study period not less than 120 days after chemotherapy or the last dose of toripalimab (whichever is later).

Exclusion Criteria:

1. Patients with lung adenocarcinoma with confirmed EGFR mutations or ALK rearrangements;
2. Histological evidence of small cell components;
3. Patients with other malignant tumors within five years prior to the start of this trial;
4. Having received any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment, and experimental treatment, etc.;
5. Concomitant unstable systemic diseases, including active infections, uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg), unstable angina, angina that started within the last 3 months, congestive heart failure (≥New York Heart Association [NYHA] Class II), myocardial infarction (within 6 months prior to enrollment), severe arrhythmias requiring drug treatment, liver, kidney, or metabolic diseases;
6. Active, known, or suspected autoimmune diseases, or autoimmune paraneoplastic syndromes requiring systemic treatment;
7. Allergy to the trial drug;
8. Currently diagnosed with interstitial lung disease;
9. Concomitant HIV infection or active hepatitis;
10. Pregnant or lactating women;
11. Patients with neurological or psychiatric disorders who are unable to cooperate;
12. Concurrently participating in another therapeutic clinical study;
13. Other situations deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) rate | Up to 30 months
  PCR rate is defined as the proportion of participants who have achieved pathologic complete response (on routine hematoxylin and eosin staining, no tumor cell can be found in tumor bed or lymph node) in all participants.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 60 months
  Event-free survival (EFS) is defined as the length of time (months) from randomization to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause. Participants who don't undergo surgery for reason other than progression will be considered to have an event at progression or death. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Overall survival (OS) | Up to 60 months
  It is defined as the time (months) from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Major pathologic response (MPR) rate | Up to 30 months
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants.
Objective response rate (ORR) | Up to 30 months
  ORR is defined according to the RECIST v1.1 criteria.
R0 resection rate | Up to 30 months
  R0 resection rate is defined as the proportion of participants who have achieved R0 resection (complete resection with no residual tumor cell in the resection margin) in all participants.
Treatment-related adverse event (TRAE) | Up to 30 months
  TRAE is defined and classified according to NCI-CTCAE v5.0 in all participants.
Health related quality of life (HRQol) composite | Up to 5 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.